CLINICAL TRIAL: NCT00759369
Title: Water as Therapy in Autosomal Dominant Polycystic Kidney Disease
Brief Title: Water as Therapy in Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11451
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Water prescription
  Interventions: Other: Water prescription

INTERVENTIONS:
Other: Water prescription — Water prescription in 12 to 16 equally divided doses

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is the most common single gene disorder that is potentially fatal. ADPKD is caused by mutations in either of two genes (PKD1, PKD2). Cysts begin to develop primarily in renal collecting tubules in utero and continue to form and expand throughout the patient's life. One of the goals of the study is to formulate a water prescription for use in clinical trials to determine the effect of sustained water diuresis on the progression of ADPKD.

DETAILED DESCRIPTION:
The proposed study will devise a quantitative model to estimate the amount of water an individual would need to ingest in order to lower the 24 h mean urine osmolality to a level below plasma (~285 mOsm/Kg). This osmolality goal is chosen because the 24h median urine osmolality of humans is ordinarily ~753 mOsm/Kg, much greater than 285 mosm/Kg (6, 7). In other words, normal humans are usually anti-diuretic during waking hours and while asleep. Median 24h urine volume is ~1225 ml (range 1051 - 2270). In temperate climates the insensible losses of water in sweat, respiration and stool are nearly balanced by the water ingested in solid and semi-solid foods and derived from metabolism. Thus, daily urine volume measured upon arising in the morning is a reasonably good indicator of the volume of fluids drunk over the preceding 24 h.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD verified by ultrasound, CT or MRI, family history or physical exam
* Normal creatinine clearance, calculated by Cockroft-Gault formulat
* Good general health
* Controlled blood pressure, < 140/90
* Absence of urinary tract symptoms such as dysuria, hesitancy, diminished flow

Exclusion Criteria:

* Azotemia
* Uncontrolled hypertension
* Urinary tract symptoms, dysuria, hesitancy, diminished flow, gross hematuria
* Diabetes mellitus, cancer, hematologic disorder
* Unable to follow directions
* Solitary kidney
* History of CHF, liver dysfunction or hyponatremia
* Currently taking diuretics
* Nephrotic range proteinuria (3.5 g/day)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Percentage of mean urine osmolality decreased from baseline | Day 3, 4, 5

SECONDARY OUTCOMES:
Number of individuals who have an average daily solute excretion within 16.5% of baseline | End of study
Number of individuals whose average total urine volume is within 18% of baseline. | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Connie Wang, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Wang CJ, Creed C, Winklhofer FT, Grantham JJ. Water prescription in autosomal dominant polycystic kidney disease: a pilot study. Clin J Am Soc Nephrol. 2011 Jan;6(1):192-7. doi: 10.2215/CJN.03950510. Epub 2010 Sep 28. PMID 20876670